CLINICAL TRIAL: NCT04635137
Title: Percutaneous Ablation and Cementoplasty for Painful Bone Lesions: A Canadian Single-Centre Experience
Brief Title: Ablation and Cementoplasty for Painful Bone Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Jason Wong, Interventional Radiologist; Clinical Associate Professor, University of Calgary, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB20-1593
Record Dates: First submitted 2020-11-09; First posted 2020-11-18 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Bone Lesion; Bone Metastases; Spine Metastases
Keywords: Ablation; Cementoplasty; Pain Palliation
MeSH Terms: interventions — Cementoplasty

STUDY DESIGN:
Intervention Model Description: Single-arm prospective study of pain and quality of life before and after ablation/cementoplasty procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation and Cementoplasty (Experimental): All patients undergoing thermal ablation and cementoplasty procedure for one or more painful bone lesion
  Interventions: Procedure: Ablation and Cementoplasty

INTERVENTIONS:
Procedure: Ablation and Cementoplasty — Percutaneous thermal ablation with subsequent cementoplasty in a single procedure

SUMMARY:
The aim of this research study is to assess the effectiveness of combined ablation and cementoplasty in the treatment of spinal, pelvic, and extraspinal lesions causing pain resistant to conventional treatment at our centre. In particular, the investigator seek to verify the safety and efficacy for multiple primary tumor types and benign lesions as well as encompass multiple measurements of outcome, including visual analog scale (VAS) for pain, opioid and analgesic use, and overall performance scales, combined with cross-sectional imaging follow-up to assess tumor burden, to ascertain a comprehensive Canadian single-centre experience that has been lacking in previous studies.

DETAILED DESCRIPTION:
Research Question & Objectives

1. To conduct a prospective, single-centre study of combined ablation and cementoplasty treatment for painful spinal and extraspinal osseous lesions.
2. Report the technical outcome and safety of percutaneous ablation prior to image-guided cementoplasty in a single treatment session.
3. Review the effectiveness and durability of pain control, local tumor control, and the impact on QoL using ablation and cementoplasty in treating spinal/extraspinal osseous tumors.
4. Assess the feasibility and efficacy of ablation and cementoplasty treatment for different primary tumor types and benign lesions.

Research Design

The investigators will conduct a single-centre, single-arm, cohort analysis of all patients who undergo cementoplasty for osseous disease in the department of interventional radiology over a two-year period. This will be a prospective paired comparison study with patients serving as their own controls. Technical success and procedural complications will be monitored and recorded for all patients. All patients will be followed until death or 3 months post-procedure.

The investigators aim to enroll a minimum of 40 patients referred for symptomatic osseous lesions. Bipolar radiofrequency ablation (Osteocool RFA system, Medtronic) or cryoablation (Visual Ice Cryoablation, Boston Scientific) will be performed under CT, ultrasound, or fluoroscopic guidance at the discretion of the treating radiologist, and immediately followed by cement injection. Radiological outcomes, including local tumor control and disease progression, will be assessed by CT imaging immediately post-procedure as well as 3-month follow-up. Clinical outcomes will be evaluated by VAS, analgesic use, and QoL assessment using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) prior to procedure and immediately post-procedure, as well at 1-week, 1-month, and 3-month intervals post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* adult patient with spinal, pelvic, or extraspinal bone lesion
* pain clinically localized to a single region and tumor involvement confirmed with imaging
* life expectancy greater than 3 months
* provision of informed consent

Exclusion Criteria:

* non-correctable coagulation disorder
* systemic or localized infection
* multiple painful lesions requiring different treatment approaches
* neurological deficits or radicular neurological symptoms
* rheumatic disease
* pregnancy
* previous ablation and/or cementoplasty treatment to same lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Pain Scale | Pre-procedure
  Visual Analog Scale; values 0-10 with 0 being no pain and 10 being the worst pain imaginable.
Pain Scale | immediately post-procedure
  Visual Analog Scale; values 0-10 with 0 being no pain and 10 being the worst pain imaginable.
Pain Scale | 1 week post-procedure
  Visual Analog Scale; values 0-10 with 0 being no pain and 10 being the worst pain imaginable.
Pain Scale | 1 month post-procedure
  Visual Analog Scale; values 0-10 with 0 being no pain and 10 being the worst pain imaginable.
Pain Scale | 3 months post-procedure
  Visual Analog Scale; values 0-10 with 0 being no pain and 10 being the worst pain imaginable.
Quality of Life Questionnaire | Pre-procedure
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). The QLQ-C30 is composed of 3 multi-item scales including a functional scale, a global health status/quality of life scale, and a symptom scale. Each scale ranges in score from 0-100 with a higher scale score representing a high/healthy level of functioning, quality of life, and symptomatology/problems, respectively.
Quality of Life Questionnaire | immediately post-procedure
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). The QLQ-C30 is composed of 3 multi-item scales including a functional scale, a global health status/quality of life scale, and a symptom scale. Each scale ranges in score from 0-100 with a higher scale score representing a high/healthy level of functioning, quality of life, and symptomatology/problems, respectively.
Quality of Life Questionnaire | 1 week post-procedure
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). The QLQ-C30 is composed of 3 multi-item scales including a functional scale, a global health status/quality of life scale, and a symptom scale. Each scale ranges in score from 0-100 with a higher scale score representing a high/healthy level of functioning, quality of life, and symptomatology/problems, respectively.
Quality of Life Questionnaire | 1 month post-procedure
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). The QLQ-C30 is composed of 3 multi-item scales including a functional scale, a global health status/quality of life scale, and a symptom scale. Each scale ranges in score from 0-100 with a higher scale score representing a high/healthy level of functioning, quality of life, and symptomatology/problems, respectively.
Quality of Life Questionnaire | 3 months post-procedure
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). The QLQ-C30 is composed of 3 multi-item scales including a functional scale, a global health status/quality of life scale, and a symptom scale. Each scale ranges in score from 0-100 with a higher scale score representing a high/healthy level of functioning, quality of life, and symptomatology/problems, respectively.
Analgesia | Pre-procedure
  Opioid and non-opioid analgesia use
Analgesia | immediately post-procedure
  Opioid and non-opioid analgesia use
Analgesia | 1 week post-procedure
  Opioid and non-opioid analgesia use
Analgesia | 1 month post-procedure
  Opioid and non-opioid analgesia use
Analgesia | 3 months post-procedure
  Opioid and non-opioid analgesia use

SECONDARY OUTCOMES:
Disease Burden | 3 months post-procedure
  Tumor burden as assessed by CT scan following procedure as compared to pre-procedure scan

CONTACTS AND LOCATIONS:
Overall Officials: Jason K Wong, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - South Health Campus, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: No